CLINICAL TRIAL: NCT07092241
Title: The Efficacy of Beneficial Intestinal Microbiota in the Treatment of Migraine and Its Mechanism: Basic and Clinical Studies
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202207086RIND
Record Dates: First submitted 2025-07-08; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Migraine
Keywords: pediatric migraine; gut-brain-axis
MeSH Terms: interventions — Microbiota

STUDY DESIGN:
Intervention Model Description: Double set parallel
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The placebo group (Placebo Comparator): Double set parallel
  Interventions: Dietary Supplement: microbiota
- treated group (Active Comparator)
  Interventions: Dietary Supplement: microbiota

INTERVENTIONS:
Dietary Supplement: microbiota — Bifidobacterium breve and Bifidobacterium longum
Dietary Supplement: microbiota — Bifidobacterium and Lactobacillus
  Arms: The placebo group

SUMMARY:
pediatric migraine

DETAILED DESCRIPTION:
To explore the efficacy and pathogenesis of gut-brain axis by basic and clinical approach, The investigators will apply the candidate beneficial bacteria selected from the results of our previous clinical studies to the migraine animal model and will further conduct a clinical trial that investigates the efficacy of the commercial probiotics containing these candidate beneficial bacteria for the pediatric migraineurs to explore their therapeutic potential in treating migraine. The participants will keep headache diary and disability assessment by Pediatric Migraine Disability Assessment Score (PedMIDAS: 0-240) will be evaluated before and at the end of 12 weeks therapy. The investigators will also examine the effects of the protective bacteria clinically by measuring CGRP, a key biomarker of migraine, and proinflammatory cytokines before and after treatment by clinical approach, and explore these important markers on both the gut and brain ends in the migraine animal model to clarify the mechanism of gut-brain axis in migraine pathogenesis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis with migraine

Exclusion Criteria:

1. Receiving antibiotic treatment for the past 2 weeks
2. Receiving probiotic treatment for the past one month
3. Multiple congenital anomalies, for instance, meningoencephalocele, chromosomal anomalies, and congenital intestinal atresia, etc.
4. Mental retardation that is difficult to describe the symptoms

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The efficacy of beneficial intestinal microbiota in the treatment of migraine and its mechanism: basic and clinical studies | From enrollment to the end of treatment at 12 weeks
  evaluation of the efficacy: headache intensity (pain score: 0-10), frequency (headache times per week) and headache days per week as well as disability assessment by Pediatric Migraine Disability Assessment Score (PedMIDAS: 0-240). The listed outcome measures are all distinct clinical assessments related to migraine burden and are not derived from or dependent on variables such as weight or height. Each outcome is measured using its own standardized scale or unit and will be reported separately as specified in the protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data will not be shared due to privacy concerns and the lack of participant consent for public data sharing. Additionally, the scope of the study does not include provisions for data sharing beyond the primary analyses.